CLINICAL TRIAL: NCT04202874
Title: A Double-blinded Randomized Trial Comparing Surgeon-administered Transversus Abdominis Plane (TAP) Block With Placebo After Midline Laparotomy in Gynecologic Oncology
Brief Title: A Trial Comparing Surgeon-administered TAP Block With Placebo After Midline Laparotomy in Gynecologic Oncology
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Laurence Bernard, Fellow, Gynecology Oncology, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8302
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Genital Neoplasm Malignant Female; Surgical Procedure, Unspecified
Keywords: randomized controlled trial; Transversus Abdominis Plane block

STUDY DESIGN:
Intervention Model Description: Eighty women above the age of 18 and undergoing a midline laparotomy for a suspected gynecologic malignancy will be randomized to undergo a bilateral surgeon-administered Tranversus abdomens plane block with either 40ml of 0.25% bupivacaine or an equal volume of saline administered equally over both sides (placebo), prior to fascial closure. Forty patient will receive bupivacaine, and 40 patients will receive the placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient, surgeon, anesthesiologist, scrub nurse and outcome assessors will be blinded. The operating room circulating nurse, who will be providing the substance, will be unblinded. The investigators will be unblinded after data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine (Experimental): Administration of 20ml of bupivacaine 0.25% on each side, for a total of 40ml.
  Interventions: Procedure: Surgeon-administered transversus abdominis plane (TAP)
- Saline (Placebo Comparator): Administration on 20ml of normal saline on each side, for a total of 40ml.
  Interventions: Procedure: Surgeon-administered transversus abdominis plane (TAP)

INTERVENTIONS:
Procedure: Surgeon-administered transversus abdominis plane (TAP) — Prior to fascial closure, the rectus muscle is gently elevated superiorly and the surgeon identifies its lateral border; the nerves that supply the anterior abdominal wall travel through the myofascial plane between internal oblique and transversus abdominis muscles, 2 fingerbreadths above the iliac crest. Access to this plane can easily be achieved by inserting a blunted needle through the parietal peritoneum; there is an appreciable loss of resistance ('one pop') and the correct plane is entered. After careful aspiration to ensure no vascular injury has occurred, 20 mL 0.25% bupivacaine or 20 mL of normal saline is injected slowly. The same procedure is repeated on the other side.

SUMMARY:
Multimodal opioid-sparing analgesia is recommended in order to prevent post-operative complications and shorten length of stay. Administration by the surgeon of local anesthetics in the abdominal wall after surgery for a suspected gynaecological malignancy will be studied. Eighty women above the age of 18 and undergoing a midline laparotomy for a suspected gynecologic malignancy will be recruited. Half of these women will received a Transversus Abdominis Plane (TAP) block using local anesthetics, and half will receive a placebo (saline water). The primary outcome studied will be the total dose of opioid in morphine equivalents received in the postoperative period. The primary hypothesis is that surgeon-performed TAP blocks reduce the need for opioids after surgery. Secondary outcomes including postoperative pain scores, postoperative nausea and vomiting rates, time to flatus, incidence of clinical ileus and time to discharge from hospital will also be recorded.

DETAILED DESCRIPTION:
Multimodal opioid-sparing analgesia is recommended in order to prevent post-operative complications and shorten length of stay. While ultrasound-guided Transversus Abdominis Plane (TAP) block has been shown to reduce postoperative opioid use, the time and expertise needed to perform it can be a barrier to administering the procedure. A surgeon-administered TAP block has been described, but has yet to be evaluated with a randomized controlled study in gynecology oncology patients undergoing a midline laparotomy. The investigators hypothesize that surgeon-administered TAP blocks may decrease total opioid use in the first 24 hours.

Eighty women above the age of 18 and undergoing a midline laparotomy for a suspected gynecologic malignancy will be recruited to undergo bilateral surgeon-administered TAP blocks with either 40ml of 0.25% bupivacaine or an equal volume of saline administered equally over both sides, prior to fascial closure. Exclusion criteria include inability to give informed consent, presence of contraindications or sensitivities to drugs specified in the protocol, pre-existing truncal sensory disturbance, history of chronic opioid use, infections at the injection site, significant adhesions on the anterior or lateral abdominal wall preventing access to the injection site, patients receiving neuraxial anesthesia (Epidural, Spinal) or local wound infiltration. The primary outcome studied will be the total dose of opioid in morphine equivalents received in the postoperative period. Secondary outcomes including postoperative pain scores, postoperative nausea and vomiting rates, time to flatus, incidence of clinical ileus and time to discharge from hospital will also be recorded.

Sample size calculation was based on a meta-analysis by Johns for use of TAP blocks in abdominal surgeries, that reported morphine equivalents mean at 24h as 20.6mg for the TAP group and 44.3mg for the control group (mean difference of 23mg in 24h), with a standard deviation of 14mg. To find a clinically significant decrease in opioid use of 20%, our primary outcome, with a 2-tailed analysis and power of 80%; the investigators would need 36 patients in each group. To account for potential dropouts and protocol violations, as well as secondary analyses, the investigators will recruit a total of 80 patients (40 in the TAP block group and 40 controls).

Differences in characteristics between treatment and control groups will be analysed using the chi-square test for dichotomous data, independent samples Student's t-test for parametric continuous variables, and Mann-Whitney U test for non-parametric continuous data. Test of normality will be performed using the Shapiro-Wilk test. If there is significant (>10%) missing data, data will be imputed by predictive mean matching. Subgroup analysis by type of incision (infraumbilical vs supraumbilical) will be performed.

Missing data and patterns will be assessed monthly by the data manager. Remedial measures, including retraining of staff, will be used as needed to minimize missing data. The investigators plan for an intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above undergoing elective gynecologic oncology surgery for a suspected malignancy using a midline laparotomy incision.

Exclusion Criteria:

1. Patients unable to give informed consent
2. Patients with contraindications or sensitivities to drugs specified in the protocol
3. Pre-existing truncal sensory disturbance
4. History of chronic opioid use (daily use > 3 months)
5. Infections at the injection site
6. Significant adhesions on the anterior abdominal wall preventing access to the injection site
7. Concurrent, non-abdominal surgical procedure performed at the same time
8. Patients receiving neuraxial anesthesia/analgesia (epidural, spinal) or local wound infiltration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Total dose of opioid (in morphine equivalents) received in the postoperative period | 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative pain scores | at 4, 8, 12, 16, 20, 24, 30, 36, 42 and 48 hours after surgery
  Numerical Pain Rating Scale, from 0 to 10. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Postoperative nausea and vomiting rates | postoperative day 1
  As defined by the Simplified Postoperative Nausea and Vomiting (PONV) impact scale
Time to flatus | During admission
  In hours
Incidence of clinical ileus | During admission
  as a surgeon's diagnosis of postoperative ileum, including diagnosis on abdominal x-ray, return to nothing-by-mouth status, or (re)insertion of a nasogastric tube.
Time to discharge from hospital | During admission
  In hours

CONTACTS AND LOCATIONS:
Overall Officials: Clare Reade, MD, Principal Investigator — McMaster University
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] McDermott G, Korba E, Mata U, Jaigirdar M, Narayanan N, Boylan J, Conlon N. Should we stop doing blind transversus abdominis plane blocks? Br J Anaesth. 2012 Mar;108(3):499-502. doi: 10.1093/bja/aer422. Epub 2012 Jan 11. PMID 22236911
- [Background] Owen DJ, Harrod I, Ford J, Luckas M, Gudimetla V. The surgical transversus abdominis plane block--a novel approach for performing an established technique. BJOG. 2011 Jan;118(1):24-7. doi: 10.1111/j.1471-0528.2010.02779.x. Epub 2010 Nov 18. PMID 21083866
- [Background] Ravichandran NT, Sistla SC, Kundra P, Ali SM, Dhanapal B, Galidevara I. Laparoscopic-assisted Tranversus Abdominis Plane (TAP) Block Versus Ultrasonography-guided Transversus Abdominis Plane Block in Postlaparoscopic Cholecystectomy Pain Relief: Randomized Controlled Trial. Surg Laparosc Endosc Percutan Tech. 2017 Aug;27(4):228-232. doi: 10.1097/SLE.0000000000000405. PMID 28472015
- [Background] Baeriswyl M, Kirkham KR, Kern C, Albrecht E. The Analgesic Efficacy of Ultrasound-Guided Transversus Abdominis Plane Block in Adult Patients: A Meta-Analysis. Anesth Analg. 2015 Dec;121(6):1640-54. doi: 10.1213/ANE.0000000000000967. PMID 26397443
- [Background] Charlton S, Cyna AM, Middleton P, Griffiths JD. Perioperative transversus abdominis plane (TAP) blocks for analgesia after abdominal surgery. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD007705. doi: 10.1002/14651858.CD007705.pub2. PMID 21154380
- [Background] Johns N, O'Neill S, Ventham NT, Barron F, Brady RR, Daniel T. Clinical effectiveness of transversus abdominis plane (TAP) block in abdominal surgery: a systematic review and meta-analysis. Colorectal Dis. 2012 Oct;14(10):e635-42. doi: 10.1111/j.1463-1318.2012.03104.x. PMID 22632762
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Chang H, Rimel BJ, Li AJ, Cass I, Karlan BY, Walsh C. Ultrasound guided transversus abdominis plane (TAP) block utilization in multimodal pain management after open gynecologic surgery. Gynecol Oncol Rep. 2018 Oct 15;26:75-77. doi: 10.1016/j.gore.2018.10.007. eCollection 2018 Nov. PMID 30364775
- [Background] Narasimhulu DM, Scharfman L, Minkoff H, George B, Homel P, Tyagaraj K. A randomized trial comparing surgeon-administered intraoperative transversus abdominis plane block with anesthesiologist-administered transcutaneous block. Int J Obstet Anesth. 2018 Aug;35:26-32. doi: 10.1016/j.ijoa.2018.04.007. Epub 2018 Apr 27. PMID 29914782
- [Background] Chandrakantan A, Glass PS. Multimodal therapies for postoperative nausea and vomiting, and pain. Br J Anaesth. 2011 Dec;107 Suppl 1:i27-40. doi: 10.1093/bja/aer358. PMID 22156268
- [Background] Kaye AD, Urman RD, Rappaport Y, Siddaiah H, Cornett EM, Belani K, Salinas OJ, Fox CJ. Multimodal analgesia as an essential part of enhanced recovery protocols in the ambulatory settings. J Anaesthesiol Clin Pharmacol. 2019 Apr;35(Suppl 1):S40-S45. doi: 10.4103/joacp.JOACP_51_18. PMID 31142958
- [Background] Bakkum-Gamez JN, Langstraat CL, Martin JR, Lemens MA, Weaver AL, Allensworth S, Dowdy SC, Cliby WA, Gostout BS, Podratz KC. Incidence of and risk factors for postoperative ileus in women undergoing primary staging and debulking for epithelial ovarian carcinoma. Gynecol Oncol. 2012 Jun;125(3):614-20. doi: 10.1016/j.ygyno.2012.02.027. Epub 2012 Feb 24. PMID 22370599
- [Derived] Bernard L, Lavecchia M, Trepanier G, Mah S, Pokoradi A, McGinnis JM, Alyafi M, Glezerson B, Nguyen J, Carlson V, Helpman L, Elit L, Jimenez W, Eiriksson L, Reade CJ. A double-blinded, randomized trial comparing surgeon-administered transversus abdominis plane block with placebo after midline laparotomy in gynecologic oncology surgery. Am J Obstet Gynecol. 2023 May;228(5):553.e1-553.e8. doi: 10.1016/j.ajog.2023.02.010. Epub 2023 Feb 14. PMID 36791986